CLINICAL TRIAL: NCT00096837
Title: An Open-Label Phase II Trial of Motexafin Gadolinium (MGd) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Motexafin Gadolinium for the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0215
Record Dates: First submitted 2004-11-16; First posted 2004-11-17 (Estimated); Last update posted 2006-06-08 (Estimated); Status verified 2006-06

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium Injection

SUMMARY:
The purpose of the study is to determine if the drug motexafin gadolinium will be an effective treatment for patients who have relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or Refractory Multiple Myeloma
* ≥ 18 years old
* Able to provide consent for participation
* ECOG status 0-2

Lab values:

* ANC ≥ 1,000/µL
* WBC count ≥ 2.0/µL
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 50,000/µL
* AST and ALT ≤ 2 x ULN
* Total Bilirubin ≤ 2 x ULN
* Creatinine ≤ 2.0 mg/dL

and

* Not pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25

PRIMARY OUTCOMES:
Rate of complete response, partial response and stable disease (clinical benefit rate)

SECONDARY OUTCOMES:
Progression-free survival
Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois, United States